CLINICAL TRIAL: NCT06570590
Title: A Prospective Study of the Minimally Invasive Lapidus Procedure for Hallux Valgus Deformities Randomized With Arthroscopy or No Arthroscopy at St. Paul's Hospital in Vancouver, Canada
Brief Title: Prospective Study of Minimally Invasive Lapidus Procedure for Hallux Valgus Deformities
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Paul's Hospital, Canada (Other)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Principal Investigator, Alastair Younger, Orthopaedic Surgeon, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H23-03971
Record Dates: First submitted 2024-05-14; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Hallux Valgus and Bunion
MeSH Terms: conditions — Hallux Valgus; Bunion | interventions — Arthroscopy

STUDY DESIGN:
Intervention Model Description: 58 patients total. 29 will be randomly assigned to arthroscopy group, 29 will be randomly assigned to mini open group.
Masking Description: Patients find out their assignment group after their surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Arthroscopy (Active Comparator): Using arthroscopy in minimally invasive lapidus procedure is the current standard of care. However a new screw is used (PROstep MIS 5mm Chamfer Screw). The new hardware is expected to be substantially equivalent to standard of care.
  Interventions: Procedure: Minimally invasive lapidus procedure with arthroscopy
- No Arthroscopy (Experimental): Non-Arthroscopic Mini Arthrotomy Procedure (research-specific): Surgical procedure between the two treatment groups are equivalent except at the step of checking cartilage removal. After use of the cartilage burr the surgeon will make a small dorsal portal and use this to ensure that the cartilage is removed and all debris removed. The incision will be 2 cm long and centered over the dorsal medial aspect of the joint. The Principal Investigator wants to know if the mini arthrotomy procedure is as effective as the control because this procedure is faster and easier to perform.
  Interventions: Procedure: Minimally invasive lapidus procedure with no arthroscopy

INTERVENTIONS:
Procedure: Minimally invasive lapidus procedure with no arthroscopy — The two procedures, with and without arthroscopy, only differ by the method of assessing cartilage removal. Cartilage removal will be assessed arthroscopically in the procedure with arthroscopy. In the procedure without arthroscopy, cartilage removal will be assessed via direct visualization through a mini arthrotomy procedure. After use of the cartilage burr the surgeon will make a small dorsal portal and use this opening to ensure that the cartilage is removed and all debris removed. The incision will be 2 cm long and centered over the dorsal medial aspect of the joint.
  Other Names: No arthroscopy; MIS no arthroscopy; mini arthrotomy
  Arms: No Arthroscopy
Procedure: Minimally invasive lapidus procedure with arthroscopy — After removal of the cartilage with the cartilage burr, a 3.0 arthroscope will be inserted to inspect the joint for all cartilage removal. Any residual cartilage pieces will be removed to ensure complete cartilage debridement from the subchondral bone and fragments removed from the joint.
  Other Names: With scope
  Arms: Arthroscopy

SUMMARY:
The Lapidus procedure corrects bunions, a condition called hallux first ray deformity. Using minimally invasive surgery (MIS) to perform this procedure on patients with hallux valgus deformity is a newer approach. Because it's newer, there is not studies on how patients feel about it directly through patient reported outcomes (PROMs), which involve patients filling out questionnaires. Previous studies have looked at information that could be gathered from radiographs. This study looks specifically at how well bones heal after the MIS procedure and how patients feel about it based on their recorded responses in PROMs. The Lapidus procedure involves a step where the surgeon checks for the amount of cartilage removal, which can be done by inserting a mini camera into the joint (arthroscopically) or through a small incision for visual inspection. These two methods of checking cartilage removal are the two treatment groups for this study that patients are randomly assigned to.

The main goals of the study are as follows:

* To determine healing in minimally invasive Lapidus. Evaluated by bones fusing together at 12 weeks post-operation.
* To determine patient reported outcomes following Lapidus procedures
* To determine the relationship between patient-reported outcomes and percent bone healing.
* To assess the nonunion (bone not fusing together) rate and re-operation rate following Lapidus procedures
* To assess the correction achieved on radiographic and standing CT measurements.
* To compare radiographic and Standing CT assessment of hallux valgus deformity and correction after surgery.

ELIGIBILITY:
Inclusion Criteria:

* The subject is at least 19 years of age.
* The subject is considered to be skeletally mature.
* The subject is undergoing an isolated 1st TMT, which may or may not include concomitant procedures, such as:

  * Soft tissue realignment
  * Heel cord lengthening
  * Akin osteotomy
  * Lesser toe osteotomies or claw toe correction
* The subject is able to comply with all post-operative evaluations and visits.
* The subject is able to provide informed consent.
* The subject consents to and will receive either arthroscopy or no arthroscopy condition using the PROstep MIS 5mm Chamfer Screw.

Exclusion Criteria:

* Patients indicated for TMT fusion for non-hallux valgus procedures.
* Patients with simultaneous fusion of second and third ray.
* Patients indicated for navicular-cuneiform joint performed at the same time.
* The subject has:

  * Arthritis in the affected joint
  * Severe osteoporosis
  * Neuromuscular impairment
  * Prior or current infection in the affected joint
  * Charcot foot
* The subject has undergone previous fusion surgery of the proposed site (i.e., revision of failed fusion attempt).
* The subject will be undergoing an ankle replacement, any other concomitant fusion(s), or any lesser metatarsal osteotomies in the affected foot or ankle in the same sitting.
* The subject has concomitant injury, which in the opinion of the Investigator, is likely to impair functions for as long as or longer than the recovery from the subject's 1st TMT fusion.
* The subject is deemed morbidly obese (BMI > 50 kg/m2
* The subject has a major risk factor for non-union (ex. poorly controlled diabetes, current smoker).
* There is radiographic evidence of bone cysts, segmental defects or growth plate fracture around the fusion site that may negatively impact bony fusion. The patient currently has untreated malignant neoplasm(s), or is currently undergoing radio- or chemotherapy or has been diagnosed with hypercalcemia.
* The subject is known to be pregnant during the study period.
* The Investigator judges the subject to be unable or unlikely to remain compliant to follow-up due to a physical or mental condition (ex. currently being treated for a psychiatric disorder, senile dementia, Alzheimer's disease, etc.).
* The subject is unable to provide informed consent.
* The subject is unable to communicate with the research team.
* The subject is unable to comply with follow-up.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Primary: Bone Fusion | At 12 weeks post-operation
  Rate of bone fusion by comparing the mean percentage of the joint fused at Week 12 using LineUp scans

SECONDARY OUTCOMES:
Secondary: Questionnaires-Musculoskeletal Outcomes Data Evaluation and Management System (MODEMS) | Pre-operative, and at all post-operative followups (2 Weeks, 6 Weeks, 12 Weeks, 52 Weeks)
  Patient reported outcomes as measured by MODEMS (includes AOS and SF-36) compared to baseline questionnaire.
Secondary: Questionnaires-Foot and Ankle Ability Measure (FAAM) | Pre-operative, and at all post-operative followups (2 Weeks, 6 Weeks, 12 Weeks, 52 Weeks)
  Patient reported outcomes as measured by FAAM compared to baseline questionnaire.
Secondary: Questionnaires-Pain Catastrophizing Scale (PCS) | Pre-operative, and at all post-operative followups (2 Weeks, 6 Weeks, 12 Weeks, 52 Weeks)
  Patient reported outcomes as measured by PCS compared to baseline questionnaire.
Secondary: Re-operation and complication rates | At any point during enrolment up to 52 weeks post-operation.
  Reoperations and complications will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Alastair Younger, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided